CLINICAL TRIAL: NCT05436262
Title: Using Real-time Functional Magnetic Resonance Imaging (fMRI) Neurofeedback and Motor Imagery to Enhance Motor Timing and Precision in Cerebellar Ataxia
Brief Title: Using Real-time fMRI Neurofeedback and Motor Imagery to Enhance Motor Timing and Precision in Cerebellar Ataxia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Virginia Polytechnic Institute and State University (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00300264; R21NS125546 (NIH)
Record Dates: First submitted 2022-06-23; First posted 2022-06-29 (Actual); Results first posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-12

CONDITIONS: Cerebellar Ataxia; Spinocerebellar Ataxias; Cerebellar Degeneration
Keywords: Cerebellar Ataxia; Spinocerebellar Ataxias; Cerebellar Diseases; Neurodegenerative Diseases; Cerebellum; Gait; Balance; Movement Disorders
MeSH Terms: conditions — Cerebellar Ataxia; Spinocerebellar Ataxias; Cerebellar Diseases; Neurodegenerative Diseases; Movement Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real time neurofeedback with task and at-home finger tapping practice sessions (Experimental): Participants will undergo a real-time fMRI scan during which two distinct tasks will be performed.
  Neurofeedback treatment: During the fMRI scan, the tasks consist of:
  1. Overt finger tapping in time with a flashing cue.
  2. Motor imagery (of finger tapping).
  During overt finger tapping, feedback will consist of a slider bar that indicates tapping accuracy to target speed (1 or 4Hz). During motor imagery, neurofeedback will consist of a crosshair that flashes to indicate the success of recruiting predicted brain regions (consistent with those engaged during overt tapping).
  At-home therapy: Participants are assigned to one of two groups where participants will practice each day 17 sessions total at-home.
  Group 1: Overt finger tapping on 17 daily sessions. Participants will finger tap in time with the flashing cue.
  Interventions: Device: Real-time fMRI with neurofeedback of motor imagery
- Real time neurofeedback with task and at-home motor imagery practice sessions (Experimental): Participants will undergo a real-time fMRI scan during which two distinct tasks will be performed.
  Neurofeedback treatment: During the fMRI scan, the tasks consist of:
  1. Overt finger tapping in time with a flashing cue.
  2. Motor imagery (of finger tapping).
  During overt finger tapping, feedback will consist of a slider bar that indicates tapping accuracy to target speed (1 or 4Hz). During motor imagery, neurofeedback will consist of a crosshair that flashes to indicate the success of recruiting predicted brain regions (consistent with those engaged during overt tapping).
  At-home therapy: Participants are assigned to one of two groups where participants will practice each day 17 sessions total at-home.
  Group 2: Motor imagery only on 13 daily sessions, and overt finger tapping only on 4 daily sessions.
  Interventions: Device: Real-time fMRI with neurofeedback of motor imagery

INTERVENTIONS:
Device: Real-time fMRI with neurofeedback of motor imagery — Participants undergo a real-time fMRI scan during which they are provided feedback regarding the accuracy of their motor imagery performance.

SUMMARY:
The aim of the research is to improve motor function in people with cerebellar ataxia by using neuroimaging methods and mental imagery to "exercise" motor networks in the brain. The relevance of this research to public health is that results have the potential to reduce motor deficits associated with cerebellar atrophy, thereby enhancing the quality of life and promoting independence.

ELIGIBILITY:
Inclusion Criteria:

* 18-100 years of age
* At least 8th-grade education
* Right-handedness
* Clinical diagnosis of progressive, degenerative cerebellar ataxia by a movement disorder specialist (cerebellar ataxia of unknown etiology, and spinocerebellar ataxias with and without genetic confirmation)

Exclusion Criteria:

* History of Axis I psychiatric disorders (including alcohol and drug dependence)
* Severe or unstable medical disorder, neurological disorders, such as stroke or epilepsy
* History of head injury that resulted in a loss of consciousness greater than 5 minutes and/or neurological sequelae
* Any condition that is contraindicated for the MRI environment (e.g., metal in the body, pacemaker, claustrophobia)
* Currently pregnant
* Clinical diagnosis of multiple system atrophy (MSA) or Friedrich's ataxia (FA)
* Eligible subjects may be asked to refrain from medications that affect the central nervous system that would also make data difficult to interpret (e.g., sedatives) for an appropriate period of time prior to scanning
* Participants will be excluded if the participants do not have a home computer with internet available to complete the 3-week at-home component of the study protocol

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2023-03-14 (Actual); Primary Completion 2024-01-22 (Actual); Study Completion 2024-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cherie Marvel, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Immediately following publication. No end date.
Access Criteria: Access to trial individual participant data (IPD) can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact cmarvel1@jhmi.edu.

RESULTS

PARTICIPANT FLOW:
Groups:
- Pre-Randomization: fMRI Neurofeedback: Participants will undergo a real-time fMRI scan during which two distinct tasks will be performed.
  Neurofeedback treatment: During the fMRI scan, the tasks consist of:
  1. Overt finger tapping in time with a flashing cue.
  2. Motor imagery (of finger tapping).
  During overt finger tapping, feedback will consist of a slider bar that indicates tapping accuracy to target speed (1 or 4Hz). During motor imagery, neurofeedback will consist of a crosshair that flashes to indicate the success of recruiting predicted brain regions (consistent with those engaged during overt tapping).
- Randomization: Homework Sessions With Tapping Only (Control Group): At-home therapy: Participants are assigned to one of two groups where participants will practice each day 17 sessions total at-home.
  Group 1: Overt finger tapping on 17 daily sessions. Participants will finger tap in time with the flashing cue.
- Randomization: Homework Sessions With Imagery Only (Intervention Group): At-home therapy: Participants are assigned to one of two groups where participants will practice each day 17 sessions total at-home.
  Group 2: Motor imagery only on 13 daily sessions, and overt finger tapping only on 4 daily sessions.
Period: Pre-Randomization
Arm/Group | Pre-Randomization: fMRI Neurofeedback | Randomization: Homework Sessions With Tapping Only (Control Group) | Randomization: Homework Sessions With Imagery Only (Intervention Group)
Started | 21 | 0 | 0
Completed | 20 | 0 | 0
Not Completed | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Period: Randomization
Arm/Group | Pre-Randomization: fMRI Neurofeedback | Randomization: Homework Sessions With Tapping Only (Control Group) | Randomization: Homework Sessions With Imagery Only (Intervention Group)
Started | 0 | 11 | 9
Completed | 0 | 10 | 9
Not Completed | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All participants have cerebellar ataxia.
Groups:
- Real Time Neurofeedback With Task With At-home Practice Sessions: Participants will undergo a real-time fMRI scan during which two distinct tasks will be performed.
  Neurofeedback treatment: During the fMRI scan, the tasks consist of:
  1. Overt finger tapping in time with a flashing cue.
  2. Motor imagery (of finger tapping).
  During overt finger tapping, feedback will consist of a slider bar that indicates tapping accuracy to target speed (1 or 4Hz). During motor imagery, neurofeedback will consist of a crosshair that flashes to indicate the success of recruiting predicted brain regions (consistent with those engaged during overt tapping).
  At-home therapy: Participants are assigned to one of two groups where participants will practice each day 17 sessions total at-home.
  Group 1: Overt finger tapping on 17 daily sessions. Participants will finger tap in time with the flashing cue.
  Group 2: Imagery on 13 daily sessions, and overt tapping on 4 sessions.
Arm/Group | Real Time Neurofeedback With Task With At-home Practice Sessions
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.31 (11.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 14
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20
  United Kingdom | 1
International Cooperative Ataxia Rating Scale (ICARS) [Mean (Standard Deviation); unit: units on a scale] — ICARS is a neurological exam to assess severity of symptoms, with a total possible score of 0-100, and higher scores indicate greater symptom severity.
  units on a scale | 35.43 (19.36)
Kinesthetic and Visual Imagery Questionnaire (KVIQ) [Mean (Standard Deviation); unit: units on a scale] — Scale to assess motor imagery vividness. Scores can range from 0 - 50, with higher scores indicating more intense imagery vividness.
  units on a scale | 38.00 (9.24)

OUTCOME MEASURES:

1. Primary Outcome: Change in Overt Tapping Accuracy as Assessed by Finger Tapping to a Flashing Cue at 1Hz Speed
Description: During the MRI session, accuracy on overt tapping will be measured by the distance of the actual tapping rate vs. target rate (1Hz). Accuracy at baseline will be compared to that of final assessment, which will take place before and after neurofeedback training, respectively. The difference in accuracy between the two tests create a delta measure (i.e., fewer errors in the final vs. baseline tests). This delta accuracy will indicate the magnitude of tapping accuracy improvements. Root mean squared error (RMSE) is the measure for both the baseline and post-treatment behavioral tasks. RMSE will be based on the actual number of taps per second relative to the expected number of taps per second (e.g., 1 tap for 1Hz). Then post treatment RMSE minus baseline RMSE will determine a delta RMSE. A higher RMSE signifies greater error. For the delta measure, it is expected, lower scores reflect greater improvement on the task.
Time Frame: Baseline and MRI duration, up to 1 hour
Population: One person withdrew from the MRI portion and did not complete the task. Four additional participants were unable to complete the functional MRI task as instructed, confirmed by post-experimental questionnaires. Because these people were presumably using strategies that were not of interest to the research question, their data was excluded from analysis.
Measure: Mean (Standard Deviation); unit: taps per second
Arm/Group | Pre-Randomization: fMRI Neurofeedback
Number analyzed (Participants) | 16
taps per second | .00141488 (.007294434)

2. Primary Outcome: Change in Overt Tapping Accuracy as Assessed by Finger Tapping to a Flashing Cue at 4Hz Speed
Description: During the MRI session, accuracy on overt tapping will be measured by the distance of the actual tapping rate vs. target rate (4Hz). Accuracy at baseline will be compared to that of final assessment, which will take place before and after neurofeedback training, respectively. The difference in accuracy between the two tests create a delta measure (i.e., fewer errors in the final vs. baseline tests). This delta accuracy will indicate the magnitude of tapping accuracy improvements. Root mean squared error (RMSE) is the measure for both the baseline and post-treatment behavioral tasks. RMSE will be based on the actual number of taps per second relative to the expected number of taps per second (e.g., 1 tap for 1Hz). Then post treatment RMSE minus baseline RMSE will determine a delta RMSE. A higher RMSE signifies greater error. For the delta measure, it is expected, lower scores reflect greater improvement on the task.
Time Frame: Baseline and MRI duration, up to 1 hour
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: taps per second
Arm/Group | Pre-Randomization: fMRI Neurofeedback
Number analyzed (Participants) | 16
taps per second | .00165387 (.010581808)

3. Primary Outcome: Change in At-home Overt Tapping Accuracy as Assessed by Finger Tapping to a Flashing Cue at 1Hz Speed
Description: Accuracy at baseline will be compared to that of final assessment, which will take place before and after the 3-week at-home practice sessions, respectively. The delta measure will indicate the magnitude of tapping accuracy improvements. Groups will be compared to examine differences in delta as a function of practice condition (tapping only or imagery plus tapping). RMSE (root mean squared error) is the measure for both the baseline and post-treatment behavioral tasks. RMSE will be based on the actual number of taps per second relative to the expected number of taps per second (e.g., 1 tap for 1Hz). Then post treatment RMSE minus baseline RMSE will determine a delta RMSE. A higher RMSE signifies greater error. For the delta measure, it is expected, lower scores reflect greater improvement on the task.
Time Frame: Baseline and At-home sessions (10 minutes/day), up to 23 days
Population: Four people did not complete the MRI component as instructed, and one person in the tapping only (control group) condition did not complete the final 7 at-home exercise sessions. These 5 people were excluded from at-home data analysis (a total of 3 excluded from Tapping and 2 excluded from Imagery).
Measure: Mean (Standard Deviation); unit: taps per second
Arm/Group | Randomization: Homework Sessions With Tapping Only (Control Group) | Randomization: Homework Sessions With Imagery Only (Intervention Group)
Number analyzed (Participants) | 8 | 7
taps per second | .392919831 (.6227685278) | .200339199 (.3242518927)

4. Primary Outcome: Change in At-home Overt Tapping Accuracy as Assessed by Finger Tapping to a Flashing Cue at 4Hz Speed
Description: Accuracy at baseline will be compared to that of final assessment, which will take place before and after the 3-week at-home practice sessions, respectively. The delta measure will indicate the magnitude of tapping accuracy improvements. Groups will be compared to examine differences in delta as a function of practice condition (tapping only or imagery plus tapping). RMSE (root mean squared error) is the measure for both the baseline and post-treatment behavioral tasks. RMSE will be based on the actual number of taps per second relative to the expected number of taps per second (e.g., 4 taps for 4Hz). Then post treatment RMSE minus baseline RMSE will determine a delta RMSE. A higher RMSE signifies greater error. For the delta measure, it is expected, lower scores reflect greater improvement on the task.
Time Frame: Baseline and At-home sessions (10 minutes/day), up to 23 days
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: taps per second
Arm/Group | Randomization: Homework Sessions With Tapping Only (Control Group) | Randomization: Homework Sessions With Imagery Only (Intervention Group)
Number analyzed (Participants) | 8 | 7
taps per second | .35613192 (.7481023854) | .067492801 (.5086197309)

5. Secondary Outcome: The Correlation Between MRI BOLD During Imagery and Finger Tapping Accuracy Improvements to a Flashing Cue at 1Hz as Assessed by a Correlation Coefficient
Description: This will assess the correlation between MRI Blood Oxygen Level Dependence (BOLD) during imagery and finger tapping accuracy improvement (pre- vs. post- neurofeedback training) by a correlation coefficient. The correlation coefficient ranging from -1 to 1, where the closer the coefficient is to -1 indicates a negative association and the closer the coefficient is to 1 indicates a strong positive association.
Time Frame: MRI duration, up to 1 hour
Population: as for outcome 1
Measure: Number; unit: correlation coefficient
Arm/Group | Pre-Randomization: fMRI Neurofeedback
Number analyzed (Participants) | 16
correlation coefficient
  Left Crus II cerebellum | .850
  Right Posterior Insula | .861
  Right Inferior Frontal Gyrus | .838
  Left Posterior Insula | .842
  Left Internal Capsule | .884
  Right Ventral Caudate | .850

6. Secondary Outcome: The Correlation Between MRI BOLD and Finger Tapping Accuracy to a Flashing Cue at 4Hz as Assessed by a Correlation Coefficient
Description: as for outcome 5
Time Frame: MRI duration, up to 1 hour
Population: as for outcome 1
Measure: Number; unit: correlation coefficient
Arm/Group | Pre-Randomization: fMRI Neurofeedback
Number analyzed (Participants) | 16
correlation coefficient | .688

7. Secondary Outcome: The Correlation Between the KVIQ and Imagery Accuracy of the Flashing Cross on the MRI Task as Assessed by a Correlation Coefficient
Description: The Kinesthetic and Visual Imagery Questionnaire (KVIQ), overall score ranging from 0-100, where higher scores reflect more vivid imagery) will assess imagery vividness. This will be correlated with the image accuracy measures described in Secondary Outcome Measure 5. The correlation coefficient ranging from -1 to 1, where the closer the coefficient is to -1 indicates a negative association and the closer the coefficient is to 1 indicates a strong positive association.
Time Frame: Up to 1.5 hours
Population: as for outcome 1
Measure: Number; unit: correlation coefficient
Arm/Group | Pre-Randomization: fMRI Neurofeedback
Number analyzed (Participants) | 16
correlation coefficient | .953

8. Secondary Outcome: The Correlation Between the ICARS and Imagery Accuracy Accuracy of the Flashing Cross on the MRI Task as Assessed by a Correlation Coefficient
Description: The International Cooperative Ataxia Rating Scale (ICARS), overall score ranging from 0-100, where higher scores indicate more severe neurological impairment) will assess neurological impairments. This will be correlated with image accuracy measures described in 'Secondary Outcome Measure 5. The correlation coefficient ranging from -1 to 1, where the closer the coefficient is to -1 indicates a negative association and the closer the coefficient is to 1 indicates a strong positive association.
Time Frame: Up to 1.5 hours
Population: as for outcome 1
Measure: Number; unit: correlation coefficient
Arm/Group | Pre-Randomization: fMRI Neurofeedback
Number analyzed (Participants) | 16
correlation coefficient | -.263

ADVERSE EVENTS:
Time Frame: Up To 3 Weeks
Groups:
- Pre-Randomization: fMRI Neurofeedback: Participants will undergo a real-time fMRI scan during which distinct tasks will be performed.
  Neurofeedback treatment: During the fMRI scan, the tasks consist of:
  1. Overt finger tapping in time with a flashing cue.
  2. Motor imagery (of finger tapping).
  During overt finger tapping, feedback will consist of a slider bar that indicates tapping accuracy to target speed (1 or 4Hz). During motor imagery, neurofeedback will consist of a crosshair that flashes to indicate the success of recruiting predicted brain regions (consistent with those engaged during overt tapping).
- fMRI Neurofeedback and Homework Sessions With Tapping (Control Group): Participants will undergo a real-time fMRI scan during which two distinct tasks will be performed.
  Neurofeedback treatment: During the fMRI scan, the tasks consist of:
  Overt finger tapping in time with a flashing cue. Motor imagery (of finger tapping). During overt finger tapping, feedback will consist of a slider bar that indicates tapping accuracy to target speed (1 or 4Hz). During motor imagery, neurofeedback will consist of a crosshair that flashes to indicate the success of recruiting predicted brain regions (consistent with those engaged during overt tapping).
  At-home therapy: Participants are assigned to group where participants will practice each day 17 sessions total at-home.
  Group 1: Overt finger tapping on 17 daily sessions. Participants will finger tap in time with the flashing cue.
- fMRI Neurofeedback and Homework Sessions With Imagery (Intervention Group): Participants will undergo a real-time fMRI scan during which two distinct tasks will be performed.
  Neurofeedback treatment: During the fMRI scan, the tasks consist of:
  Overt finger tapping in time with a flashing cue. Motor imagery (of finger tapping). During overt finger tapping, feedback will consist of a slider bar that indicates tapping accuracy to target speed (1 or 4Hz). During motor imagery, neurofeedback will consist of a crosshair that flashes to indicate the success of recruiting predicted brain regions (consistent with those engaged during overt tapping).
  At-home therapy: Group 2: Motor imagery only on 13 daily sessions, and overt finger tapping only on 4 daily sessions.
Arm/Group | Pre-Randomization: fMRI Neurofeedback | fMRI Neurofeedback and Homework Sessions With Tapping (Control Group) | fMRI Neurofeedback and Homework Sessions With Imagery (Intervention Group)
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/11 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/11 | 0/9
Other Adverse Events (participants affected / at risk) | 0/21 | 0/11 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-07-21): https://cdn.clinicaltrials.gov/large-docs/62/NCT05436262/Prot_SAP_000.pdf
  • Informed Consent Form (2023-08-13): https://cdn.clinicaltrials.gov/large-docs/62/NCT05436262/ICF_001.pdf